CLINICAL TRIAL: NCT06402682
Title: Management of Esophageal Atresia With Right Aortic Arch: Is the Side of Approach Important?
Status: Recruiting | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 24-HPNCL-02
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Right Aortic Arch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Right approach
  Interventions: Procedure: Right approach
- Left approach
  Interventions: Procedure: Left approach

INTERVENTIONS:
Procedure: Right approach — Right approach of the management of esophageal atresia with a right aortic arch
  Groups: Right approach
Procedure: Left approach — Left approach of the management of esophageal atresia with a right aortic arch
  Groups: Left approach

SUMMARY:
Esophageal atresia is associated with a right aortic arch in 2 to 13% of cases. Despite previous studies, consensus on the optimal surgical approach remains lacking. This study aims to analyze the management of esophageal atresia with a right aortic arch in France over three decades, to define the most effective surgical strategy and identify associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Having been operated on for esophageal atresia and right aortic arch

Exclusion Criteria:

* NO

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients born with esophageal atresia and right aortic arch between 1990 et 2022
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative complications | During the first 40 post-operative days
  Post-operative complications after Esophageal atresia repair

SECONDARY OUTCOMES:
specific complications | During the first 40 post-operative days
  Specific complications related to esophageal atresia and right aortic arch repair. The secondary outcome assessment was based on the declaration of clinical post-operative complications on patients medical file"

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Lenval, Nice, France